CLINICAL TRIAL: NCT06774339
Title: Biomarkers and Inflammation in Solid Organ Transplantation: Relationship With Short- and Long-Term Outcomes
Acronym: Bio-Trap
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: Bio-Trap; RC-2024-2790630 (Other Grant/Funding Number: Ricerca corrente 2024-2026 - Ministero della Salute)
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Solid Organ Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The tissue study involves sampling, preservation, and experimental analysis of:
  * Blood sample
  * Routine biopsies of the transplanted organ
  * Perfusion and/or preservation fluid of the transplanted organ
  * Urine sample
  * Bronchoalveolar lavage (only for lung transplants)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, tissue-based, low-risk, non-pharmacological study that will include adult patients undergoing solid organ transplantation (heart, liver, lung, kidney) followed at the following Units of the IRCCS Azienda Ospedaliero-Universitaria di Bologna (IRCCS AOUBO):

* Heart Failure and Transplants (heart-lung)
* Internal Medicine for the Treatment of Severe Organ Failures (liver)
* Nephrology, Dialysis, and Transplantation (kidney).

DETAILED DESCRIPTION:
The aim of this study is to perform objective biological measurements of inflammation and cellular senescence (i.e., plasma profiles of cytokines, inflammatory miRNAs, circulating free DNA, extracellular vesicles), immunosenescence (i.e., circulating and tissue-based leukocyte profiles of aging), and systemic and tissue aging (i.e., epigenetic clocks) in the collected cohort. These measures may help to stratify patients at higher risk of transplant failure (graft damage) or those at higher risk of cardiovascular, renal, metabolic, neoplastic complications, or increased mortality. Additionally, the study aims to implement therapeutic or prophylactic measures based on biological stratification to prevent the progression of biological damage.

It is also important to highlight that the identification of markers of cellular senescence, immunosenescence, and epigenetic aging in the recipient could define patterns that guide more appropriate and personalized immunosuppressive treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old at the time of enrollment) who have undergone at least one of the following: Liver transplant, Kidney transplant, Heart transplant, Lung transplant during the study period.
* Informed consent acquisition.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients listed for solid organ transplantation (liver, kidney, heart, lung) at the IRCCS Azienda Ospedaliero-Universitaria di Bologna will be enrolled during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events in Heart Transplantation | 7 years
  We will assess post-heart transplant adverse events based on Primary Non-Function (PNF), Primary Graft Dysfunction (PGD), Acute Rejection, Death from any cause, Chronic Rejection, and Major Infectious Complications.
Adverse Events in Liver Transplantation | 7 years
  We will assess post-heart transplant adverse events based on Primary Non-Function (PNF), Primary Graft Dysfunction (PGD), Acute Rejection, Death from any cause, Chronic Rejection, Major Infectious Complications and Major Cardiovascular Complications (MACE)
Adverse Events in Lung Transplantation | 7 years
  We will assess post-heart transplant adverse events based on Primary Non-Function (PNF), Acute Rejection, Death from any cause, Chronic Rejection, Major Infectious Complications and Endoscopic Complications.
Adverse Events in Kidney Transplantation | 7 years
  We will assess post-heart transplant adverse events based on Primary Non-Function (PNF), Delayed Graft Function (DGF), Acute Rejection, Graft Loss, Death from any cause, Chronic Rejection, and Major Cardiovascular Complications (MACE).

CONTACTS AND LOCATIONS:
Overall Officials: Marco G Masetti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS - Azienda ospedaliero-universitaria di Bologna, Bologna, Italy